CLINICAL TRIAL: NCT05069519
Title: Implementing Personalized Exercise Prescriptions Through Mobile Health in the Elderly Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021LS024
Record Dates: First submitted 2021-09-25; First posted 2021-10-06 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Facebook Condition (Experimental): Participants assigned to this intervention will take part in personalized Facebook health education, receive a smartwatch, receive weekly health education, share sentiments on Facebook, and receive personalized feedback.
  Interventions: Behavioral: Facebook Health Education
- Smartwatch Condition (Experimental): Participants assigned to this intervention will use a Fitbit to track daily physical activity (PA), share PA data remotely, and receive personalized feedback.
  Interventions: Behavioral: Personalized Smartwatch
- Combined Condition (Experimental): Participants assigned to this condition will receive both Fitbit and Facebook health education programs, (The Smartwatch and Facebook Conditions). The investigators will also provide weekly personalized feedback, based on PA data and sentiment analysis, that have been developed in prior pilot studies.
  Interventions: Behavioral: Personalized Smartwatch; Behavioral: Facebook Health Education
- Attention Control (No Intervention): Participants assigned to the control condition will not receive any intervention. They will receive a Fitbit smartwatch, and continue with their standard care currently done in their life during the intervention period.

INTERVENTIONS:
Behavioral: Personalized Smartwatch — Participants will continue with standard care, but will receive a Fitbit and be encouraged to participate in at least 150 min. moderate-to-vigorous physical activity (5 sessions aerobic exercise, 30 min. per session; and 2 sessions of strength training) per week if their body condition allows throughout the intervention period. The previously established daily and weekly exercise prescription will be offered to participants based on their previous week Fitbit data.
  PA improvements will be tailored over time based on each participant's previous week PA and they will be encouraged to increase PA by 5-10 min/week if possible depending on specific situations. Participants will save each workout and synchronize the Fitbit PA data to its app where they only share daily data and receive weekly personalized exercise prescriptions established in pilot studies.
  Arms: Combined Condition; Smartwatch Condition
Behavioral: Facebook Health Education — Participants assigned to this condition will receive a Fitbit smartwatch, continue with standard care, but will receive health education tips developed in the investigators' previous studies from a private Facebook group in which only group members and researchers can access. Additionally, the investigators will track login counts, analyze their post activity and online sentiments via texting mining and natural language processing, and then offer weekly personalized feedback based on the data to facilitate social support
  Arms: Combined Condition; Facebook Condition

SUMMARY:
Cancer remains a vital public health concern in the U.S. Research evidence has shown that physical activity provides many physical and mental health benefits after cancer diagnosis and plays an important role in reducing all-cause, cancer-related death and cancer events in the elderly cancer survivors (CS). Adopting a physically active lifestyle may decrease cancer risks, improve cancer prognosis and quality of life.

However, most CS did not achieve recommended 150 min/week of moderate-to- vigorous physical activity (PA [MVPA]). This issue is particularly pronounced for CS in low-income areas who tend to have considerably less access to PA-conducive environments compared to urban peers. To this accord, it is imperative to promote PA in elderly CS to offer appropriate supportive care. Thus, implementing innovative PA interventions with the goal of improving their self-regulatory health behaviors in CS is paramount.

DETAILED DESCRIPTION:
Cancer remains a vital public health concern in the U.S. Research evidence has shown that physical activity provides many physical and mental health benefits after cancer diagnosis and plays an important role in reducing all-cause, cancer-related death and cancer events in the elderly cancer survivors (CS). Adopting a physically active lifestyle may decrease cancer risks, improve cancer prognosis and quality of life.

However, most CS did not achieve recommended 150 min/week of moderate-to- vigorous physical activity (PA [MVPA]). This issue is particularly pronounced for CS in low-income areas who tend to have considerably less access to PA-conducive environments compared to urban peers. To this accord, it is imperative to promote PA in elderly CS to offer appropriate supportive care. Thus, implementing innovative PA interventions with the goal of improving their self-regulatory health behaviors in CS is paramount.

One promising area of technology for increasing health behaviors is mobile health (m-health), which includes new technologies such as smartphone app, wearables, and social media in improving quality of healthcare. 6-8 Recently, researchers have applied such technologies to promote health through increased individual PA and reduced sedentary behavior in CS and some findings are promising. Despite positive findings, limitations of the preceding literature such as small samples, lacked personalized prescriptions, and lacked big data analysis are worth noting. Further, geographic environment not only affects individual's PA but is also an important pathway through which socio-economic inequalities create health disparities. Intervention impacts may be magnified in environments (e.g., urban vs. rural) stimulating more PA, with urban leading to higher PA than rural. According to Social Ecological Model, combined interventions yielded better outcomes than single level interventions. Yet, few studies examined interactive effects of the technologies on PA and other outcomes in CS, a major gap for advancing tailored intervention. In response, the primary aim of this project is to examine effects of combination of a personalized smartwatch and a Facebook health education intervention on CS' PA (daily steps) as compared to personalized Facebook only, personalized smartwatch only, and attention control conditions, over a 6-month period. This project will also determine the effects of the m-health interventions on CS' personal (e.g., daily calories, fitness, body composition, quality of life, and beliefs) and interpersonal (social support) health outcomes.

Empirical evidence also suggests a positive link between community participation and emotions (e.g., empathy and satisfaction), which may facilitate social support and subsequent sustained behavior in CS. Understanding the effect of social support and positive emotions on PA promotion is current lacking and necessary for us to explore a potential new type of intervention for healthcare outcome. With the advancement of technology, social media and apps focusing on promoting a healthy lifestyle have been increasingly used in cancer prevention and management. Further, a sentiment analysis of online patient-authored text, or retrieving information about a patient's perception, has the potential to offer new insights on the health impact of online social support and behavior, but such analysis generally requires manual annotations which can be time-consuming and costly for health professionals. To gain these new insights, health informatics approaches (e.g., text mining techniques and natural language processing [NLP] of large datasets, including sentiment analysis ) can be leveraged to examine the relationship between changes in emotions and health outcomes among online community members. This study also attempts to explore the relationships between patients' sentiments, smart watch data and other health outcomes across time.

This project attempts to examine innovative m-health interventions on CS's PA and health outcomes while offering personalized exercise prescriptions via big data analysis. If successful, it can significantly impact the development of effective and remote PA programs to promote health and protect diseases in CS. Moreover, its findings can guide health professionals and local communities to initiate such novel intervention programs with the goal of promoting PA and health in elderly CS, particularly during or post the pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Have had one or more of the cancers of interest (i.e., breast, colon, bladder, prostate, endometrium, esophagus, lung, kidney & renal pelvis, stomach)
* Complete active cancer treatment at least three months prior to enrollment, with the exception of anti- hormonal therapy
* Possess an Android or Apple smartphone
* Having a Facebook account, or are willing to make one
* Engage in some type of physical activity (PA) as assessed by PA readiness survey.

Exclusion Criteria:

* Diagnosed with stage IV cancer
* Completed primary cancer treatment (e.g., surgery, radiotherapy) less than six months ago with new cancer diagnosis or recurrence

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Change in Daily Steps | 6 Months
  Participants' 1-week daily steps will be assessed using Fitbit Charger 4. They will be instructed to wear the Fitbit on the non-dominant wrist at all times throughout the study and daily steps will be recorded. Daily steps will be measured at baseline, 3 months, and 6 months, and the difference between baseline and 6 months will be reported.
Change in Daily Calories Burned | 6 Months
  Participants' 1-week daily calories burned will be assessed using Fitbit Charger 4. They will be instructed to wear the Fitbit on the non-dominant wrist at all times throughout the study and daily steps will be recorded. Daily calories burned will be measured at baseline, 3 months, and 6 months, and the difference between baseline and 6 months will be reported.

SECONDARY OUTCOMES:
Change in Body Mass Index (BMI) | 6 Months
  Participants will self-report their height and weight which will be used to calculate BMI, which is calculated as body weight (in kg) divided by height (in cm) squared. BMI will be measured at baseline, 3 months, and 6 months, and the difference between baseline and 6 months will be reported.
Change in Physical Activity Confidence Scale Score | 6 Months
  The Physical Activity Confidence Scale will be used to assess beliefs regarding self-efficacy. Belief will be measured on a five-point Likert scale (1-5) where higher values represent greater beliefs of self-efficacy. Physical Activity Confidence will be measured at baseline, 3 months, and 6 months, and the difference between baseline and 6 months will be reported.
Change in Physical Activity Pros and Cons Scale Score | 6 Months
  The Physical Activity Pros and Cons Scale will be used to assess beliefs regarding outcome expectancy. Belief will be measured on a five-point Likert scale (1-5) where higher values represent greater beliefs of outcome expectancy. Physical Activity Pros and Cons will be measured at baseline, 3 months, and 6 months, and the difference between baseline and 6 months will be reported.
Change in Social Support Scale Score | 6 Months
  The Social Support Scale will be used to assess beliefs regarding social support. Belief will be measured on a five-point Likert scale (1-5) where higher values represent greater beliefs of social support. Social support will be measured at baseline, 3 months, and 6 months, and the difference between baseline and 6 months will be reported.
Change in Patient-Reported Outcome Measurement Information System Score | 6 Months
  The Patient-Reported Outcome Measurement Information System, a five-point Likert scale (1-5), will be used to measure quality of life via physical functioning, anxiety, and depression, where higher scores represent greater quality of life. Quality of life will be measured at baseline, 3 months, and 6 months, and the difference between baseline and 6 months will be reported.

OTHER OUTCOMES:
Change in Sentiments | 6 Months
  Participants will be encouraged to post their experiences, emotions (e.g., empathy and satisfaction), concerns, peer feedback, support and comments on their separate Facebook pages, respectively. Sentiments will be assessed at baseline, 3 months, and 6 months, and the difference between baseline and 6 months will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Zan Gao, Principal Investigator — University of Minnesota School of Kinesiology
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No